CLINICAL TRIAL: NCT06046950
Title: TrEatment Targets in Rheumatoid Arthritis: a Randomized Multi-centre, Treat to Target Strategy Trial: TETRA Study
Brief Title: TrEatment Targets in Rheumatoid Arthritis: TETRA-study
Acronym: TETRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TETRA
Record Dates: First submitted 2023-08-15; First posted 2023-09-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAS28CRP-LDA (Experimental): Arm that is allocated to strive for DAS28CRP low disease activity (LDA)
  Interventions: Other: Treatment target DAS28CRP-LDA
- SDAI-remission (Experimental): Arm that is allocated to strive for SDAI-remission
  Interventions: Other: Treatment target SDAI-remission

INTERVENTIONS:
Other: Treatment target DAS28CRP-LDA — Aiming for DAS28CRP-low disease activity
  Arms: DAS28CRP-LDA
Other: Treatment target SDAI-remission — Aiming for SDAI-remission
  Arms: SDAI-remission

SUMMARY:
There is currently no cure for rheumatoid arthritis (RA), but many treatment options are available. The central aim of RA treatment is lowering disease activity. The proactive treatment strategy called treat to target (T2T) includes measuring disease activity, setting a target and adjusting treatment accordingly until the goal is reached. T2T has proven to be superior to usual care, but there is much debate regarding the most optimal treatment measure and target. The Disease Activity Score with 28-joint counts and c-reactive protein (DAS28CRP) low-disease activity (LDA) target and the more stringent Simplified Disease Activity Index (SDAI) remission target are the best validated targets. Especially the DAS28CRP is the most commonly used in research and practice, whereas the SDAI remission target is most recommended. The European Alliance of Associations for Rheumatology (EULAR) recommends to strive for remission, whereas the American College of Rheumatology (ACR) recommends to strive for LDA. In patients with new and established RA, the (cost)effectiveness of aiming for remission compared to LDA when starting and tapering antirheumatic drugs has not been directly compared. This study therefore aims to directly compare two T2T strategies, aiming at DAS28CRP-LDA and SDAI remission, in patients with established RA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA (according to the 2010 or 1987 ACR/ EULAR classification criteria and/or clinical diagnosis)
* (Starting) use of a DMARD
* Aged 16 years or older
* At most low disease activity, operationalised as DAS28-CRP <3.5 (DAS28 CRP 2.9 cut off for low disease activity with measurement error 0.6) or SDAI <19 (SDAI 11 cut off for low disease activity with measurement error of 8). A state of low disease activity is required at inclusion, as for RA patients in moderate or high disease activity there is no equipoise on the best course of action (treatment needs to be escalated).
* Fluency of Dutch or English, both written and verbally; able to fill in questionnaires
* Provided informed consent

Exclusion Criteria:

* Clinical deep remission, operationalised as SDAI <3.3 or DAS28-CRP <2.4, and an taper attempt in the past 2 years that was discontinued due to occurrence of flare.
* Fewer than 3 DMARD treatment options left for this patient (severe difficult-to-treat or refractory RA)
* Current severe comorbidity or other serious life-shortening conditions hampering trial participation
* Inability to comply with the study protocol or to provide informed consent with regard to intervention control and measuring outcomes

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Achievement of the composite clinical/radiological remission outcome | 18 months follow-up time point
  Achievement of the composite clinical/radiological remission outcome (radiographic progression ≤1 simple erosion narrowing score (SENS), AND, ≤1 swollen joint count, and being in PASS) at 18 months.

SECONDARY OUTCOMES:
The proportion of patients having radiographic progression (defined as > 1 simple erosion narrowing score (SENS) point) in both treatment arms | 18 months follow-up
The number of swollen joints at 18 months follow-up | 18 months follow-up
The proportion of patients achieving 'patient acceptable symptom state' (PASS) | 18 months follow-up
The proportion of patients who reach the predefined target for each treatment arm (DAS28CRP-LDA or SDAI remission) | 18 months follow-up
Percentage of patients that reach LDA or remission, using DAS28CRP- and SDAI-based definitions, in each treatment arm | 18 months follow-up
Daily functioning, measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) | 18 months follow-up
  The Health Assessment Questionnaire-Disability Index (HAQ-DI) will be used to measure the impact of the rheumatoid arthritis on daily functioning. A minimum score of 0 and a maximum score of 60 can be scored. A higher score means a higher impact on daily functioning.
Quality of life (QoL) as defined by the 'EuroQol 5 Dimensions with 5 levels' (EQ5D-5L) questionnaire | 18 months follow-up
  This questionnaire assesses five dimensions of health, including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension can be answered on a 5-point scale, ranging from no problems to extreme problems/unable to. A higher score means a worse outcome.
Incidence density rates of safety ((serious) adverse events, according to CTCAE criteria version 5.0) | 18 months follow-up
Drug use of the patients, consisting of the type and volume of antirheumatic drugs (glucocorticoids, DMARDS, NSAIDs) used over the 18 months period, and at 18 months visit | 18 months follow-up
Costs associated with medical consumption as assessed with the 'Institute for Medical Technology Assessment Medical Consumption Questionnaire' (iMCQ) | 18 months follow-up
Costs associated with loss of productivity as measured bij the 'Institute of Medical Technology Assessment Productivity Cost Questionnaire (iMTA PCQ) | 18 months follow-up
  This is a short generic questionnaire that measures loss of productivity (e.g., both paid and unpaid work) due to illness or recovery.
Proportion of patients of whom the rheumatologist adhered to the local guidelines to treat the patients | 18 months follow-up
  Clinicians are encouraged to adhere to protocol upfront, and adherence is actively monitored, but treatment decisions are ultimately made using shared decision making between patients and physicians. After study completion, adherence will be assessed through a comparison of the target measurements and any changes in treatment regime made by the rheumatologists.
The incidence density rate of flares | 18 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alfons Den Broeder, MD, PhD, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Netherlands

IPD SHARING:
Plan to Share IPD: No